CLINICAL TRIAL: NCT02403050
Title: Feasibility Study to Assess the Benefit of Using Fiducial Markers for Patients Receiving Radiotherapy for Cancer of the Oesophagus
Brief Title: Feasibility Study of Fiducial Markers in Oesophageal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Other Study IDs: GN14ON144
Record Dates: First submitted 2015-03-16; First posted 2015-03-31 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Esophageal Neoplasms
Keywords: Neoplasm Staging; Radiotherapy; Fiducial Markers
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Fiducial Markers

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Fiducial Markers Prospective cohort: 2 fiducial markers (Visicoils) to be placed in the tumor area at the routine endoscopic ultrasound (EUS) appointment.
  Interventions: Device: Fiducial markers
- Retrospective cohort: Images and clinical data from a retrospective group of patients without fiducial markers

INTERVENTIONS:
Device: Fiducial markers — 2 fiducial markers (Visicoils) to be placed in the tumor area
  Groups: Fiducial Markers Prospective cohort

SUMMARY:
Currently, patients of suitable fitness with non-metastatic esophageal cancer are treated with surgery, radiotherapy or chemoradiotherapy. If treated with radio or chemoradiotherapy, a Computerised tomography (CT) scan is performed and is the dataset used for planning radiotherapy. Information from the endoscopic ultrasound (EUS), performed during routine staging, is used to help localize the tumor, as tumors of the esophagus are poorly visualised on CT. This information is subjective and dependant on the clinician performing the procedure. The tumor is described in relation to common anatomical landmarks. Interpretion of this information can lead to over-compensation when attempting to cover the tumor with a radiation field, to avoid a "miss". It is thought that using fiducial markers called Visicoils placed in or adjacent to the tumor's top and bottom extent at the time of EUS, will lead to better definition of the tumor in the planning process and hence, improvement in local tumor control, and reduction in radiotherapy dose to normal tissue.

ELIGIBILITY:
Inclusion Criteria:

* esophageal adenocarcinoma or squamous carcinoma, or undifferentiated carcinoma.
* No previous radiotherapy or chemotherapy.
* Fit for radical treatment of their cancer with reasonable lung function, Fev1 >40%, and EUS planned.
* ECOG Performance Status 0-1: 0 - Fully active, able to carry on all predisease performance without restriction 1 - Restricted in physically strenuous activity

Exclusion Criteria:

* Pregnancy or breast feeding.
* Allergy to ciprofloxacin antibiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A retrospective group of patients images without markers, will be compared to a prospective group of patients who will be imaged and treated following implantation of fiducial tumor markers.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2015-03; Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Intra- and inter-observer variability of tumor target volume (cubic centimetres) estimation | baseline (pre-radiotherapy)
  Comparison of intra- and inter-observer variability in estimation of tumor target volume (mean and standard deviation) in the prospective (fiducial markers) and retrospective (no fiducial markers) cohorts. Data will be reported using planning volumes measured in cubic centimetres.

SECONDARY OUTCOMES:
Patient survival | 6 months post radiotherapy
local recurrence of tumor | 6 months post radiotherapy
  radiological or clinical evidence of disease recurrence
Patient survival | 12 months post radiotherapy
local recurrence of tumor | 12 months post radiotherapy
  radiological or clinical evidence of disease recurrence
Patient survival | 18 months post radiotherapy
local recurrence of tumor | 18 months post radiotherapy
  radiological or clinical evidence of disease recurrence
Patient survival | 2 years post radiotherapy
local recurrence of tumor | 2 years post radiotherapy
  radiological or clinical evidence of disease recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Vivienne MacLaren, MBChB, FRCP, Principal Investigator — NHS Greater Glasgow & Clyde
Locations (1):
- Beatson Oncology Centre, Glasgow, United Kingdom